CLINICAL TRIAL: NCT00138697
Title: Kinetics, Efficacy and Safety of IVIG-L (Human Normal Intravenous Immunoglobulin for Intravenous Use) in Hypogammaglobulinemia Patients
Brief Title: Kinetics, Efficacy and Safety of IVIG-L in Hypogammaglobulinemia Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB97003 (A & B)
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Hypogammaglobulinemia
Keywords: Agammaglobulinemia; Hypogammaglobulinemia; Immunoglobulins, Intravenous
MeSH Terms: conditions — Agammaglobulinemia

INTERVENTIONS:
Drug: IVIG-L

SUMMARY:
The kinetics, efficacy and safety of a liquid intravenous immunoglobulin product, IVIG-L, were studied in patients with hypogammaglobulinemia, who are regularly treated with intravenous immunoglobulin substitution therapy.

DETAILED DESCRIPTION:
Sanquin has developed, in cooperation with the Finnish Red Cross Blood Transfusion Service (FRCBTS), a liquid intravenous immunoglobulin product, IVIG-L. The liquid formulation of intravenous immunoglobulin simplifies the infusion, eliminates possible mistakes in the reconstitution with water for injections and reduces the space requirements in storage.

In addition to the donor selection and donor screening, several viral safety steps have been included into the production process.

In this clinical trial, the efficacy and safety of IVIG-L in patients with hypogammaglobulinemia, who are regularly treated with intravenous immunoglobulin substitution therapy, will be studied. IVIG-L will also be studied in patients with chronic ITP (KB98001). Data from both studies will be used for an application for marketing authorisation in Finland and the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Primary a- or hypogammaglobulinemia, particularly patients with X-linked agammaglobulinemia (XLA) or Common Variable Immunodeficiency (CVID)
* Used to replacement treatment with intravenous immunoglobulin with 2-4 week intervals
* A stable clinical situation (no activity of any other disease; a stable immunoglobulin dose)
* Age > 18 years
* The patient/legally acceptable representative has signed the consent form

Exclusion Criteria:

* Treatment with any other investigational drug within 7 days before study entry or previous enrolment in this study
* Known allergic reactions to human plasma or plasma products
* Have an ongoing progressive terminal disease, including HIV infection
* Pregnancy or lactation
* Known insufficiency of coronary or cerebral circulation
* Have renal insufficiency (plasma creatinine > 115µmol/L)
* Have an ongoing active disease causing general symptoms, e.g. chronic active hepatitis, persistent enterovirus infection.
* Have IgA deficiency, and anti-IgA antibodies have been detected
* Active systemic lupus erythematosus (SLE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2001-05; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Kinetics of IVIG-L in patients with hypogammaglobulinemia
Efficacy of IVIG-L in patients with hypogammaglobulinemia
Safety of IVIG-L in patients with hypogammaglobulinemia

SECONDARY OUTCOMES:
To compare the IgG trough level
To compare dosage and treatment intervals

CONTACTS AND LOCATIONS:
Overall Officials: J WM van der Meer, MD, PhD, Principal Investigator — UMC St Radboud Nijmegen
Locations (6):
- Netherlands (6):
  - Medical Centre Alkmaar, Alkmaar
  - Academic Medical Centre, Amsterdam
  - Academic Hospital Groningen, Groningen
  - LUMC, Leiden
  - UMC St. Radboud, Nijmegen
  - Leyenburg Hospital, The Hague